CLINICAL TRIAL: NCT00596297
Title: Intra-Operative and Postoperative Intraocular Bleeding After Pars Plana Vitrectomy for Vitreous Hemorrhage in Diabetic Patients Previously Treated With Intravitreal Bevacizumab
Brief Title: Preoperative Bevacizumab for Vitreous Hemorrhage
Acronym: IBEVI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Daniel da Rocha Lucena, Clinics Hospital of Ribeirão Preto, School of Medicine of Riberião Preto, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBEVI; 7309/2007
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-09

CONDITIONS: Diabetic Retinopathy; Vitreous Hemorrhage
Keywords: Diabetic Retinopathy; Vitreous Hemorrhage; Bevacizumab; pars plana vitrectomy; preoperative
MeSH Terms: conditions — Diabetic Retinopathy; Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Preoperative Intravitreal bevacizumab and pars plana vitrectomy
  Interventions: Drug: bevacizumab
- B (Active Comparator): Pars plana vitrectomy only
  Interventions: Procedure: pars plana vitrectomy

INTERVENTIONS:
Drug: bevacizumab — Intravitreal bevacizumab (1.5 mg; 0,06 ml) 1 day after baseline; pars plana vitrectomy 4 weeks after baseline
  Other Names: Avastin
  Arms: A
Procedure: pars plana vitrectomy — 4 weeks after baseline
  Arms: B

SUMMARY:
The purpose of this study is to determine whether preoperative intravitreal bevacizumab is effective in reducing intra-operative and postoperative bleeding in diabetic patients submitted to pars plana vitrectomy for vitreous hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic retinopathy causing significant vitreous hemorrhage with visual acuity loss lasting more than three months in patients not previously treated and four months in those previously LASER treated.

Exclusion Criteria:

* Previous intra-ocular surgery other than cataract surgery
* Retinal detachment
* Use of anticoagulants drugs other than aspirin
* Vitreous hemorrhage clearance at week-3 study period
* History of previous thromboembolic events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Intra- and postoperative intra-ocular bleeding | 12 weeks

SECONDARY OUTCOMES:
Visual acuity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Lucena, MD, Principal Investigator — Clinics Hospital of Ribeirão Preto, School of Medicine of Ribeirão Preto, USP
Locations (1):
- Clinics Hospital of Ribeirão Preto, School of Medicine of Ribeirão Preto, USP, Ribeirão Preto, São Paulo, Brazil